CLINICAL TRIAL: NCT02232191
Title: Immunologic Response to Pneumococcal Polysaccharide Vaccine in Splenic Injury Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1036320; 51847 (Other Grant/Funding Number: Merck Investigators Study Program)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Asplenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nonoperative (Active Comparator): Pneumococcal vaccine (Pneumovax-23) will be administered within 72 hours of injury. Baseline antibody levels will be drawn at the time of vaccine administration, with response levels being drawn 4 weeks later.
  Interventions: Biological: Pneumovax-23
- Angioembolization (Active Comparator): Pneumococcal vaccine (Pneumovax-23) will be administered 14 days after embolization. Baseline antibody levels will be drawn at the time of vaccine administration, with response levels being drawn 4 weeks later.
  Interventions: Biological: Pneumovax-23
- Splenectomy (Active Comparator): Pneumococcal vaccine (Pneumovax-23) will be administered 14 days after splenectomy. Baseline antibody levels will be drawn at the time of vaccine administration, with response levels being drawn 4 weeks later.
  Interventions: Biological: Pneumovax-23

INTERVENTIONS:
Biological: Pneumovax-23

SUMMARY:
Persons without a spleen are susceptible to potentially lethal infections from certain bacteria, with pneumococcus being the most prevalent. Vaccines are provided to help protect against these infections, though they do not so with certainty. Trauma patients who sustain an injury to their spleen currently have three treatment options available for the treating surgeon - nonoperative management, embolization, or removal of the spleen. The purpose of this study is to investigate the antibody response to pneumococcal vaccine in patients undergoing these modes of therapy.

DETAILED DESCRIPTION:
The study is a multi-institutional, prospective trial, conducted primarily at the University of California, Davis Medical Center (UCDMC) by the Department of Surgery, Division of Trauma and Acute Care Surgery. The angioembolization arm will be multicenter while the nonoperative group will be enrolled only at UCDMC. There will be a total of 75 subjects, with 25 in each of the three arms (nonoperative, angioembolization, splenectomy).

Adult trauma patients (defined as those aged 18 to 65 years old) sustaining a splenic injury and planned nonoperative management, are eligible for enrollment in the nonoperative arm. The management decision for the splenic injury is entirely at the discretion of the attending trauma surgeon. Any patient who subsequently undergoes embolization or splenectomy will be withdrawn from the study.

Adult trauma patients sustaining a splenic injury and undergoing splenic artery embolization are eligible for enrollment in this arm of the study. The management decision for the splenic injury is entirely at the discretion of the attending trauma surgeon and radiologist. All patients undergoing successful splenic artery embolization (no subsequent splenectomy or splenorrhaphy, i.e., no cross-over) are eligible.

Patients managed nonoperatively will be vaccinated within three days of their diagnosis, per standard operating protocol at UCDMC. At the time of vaccination, 7cc of venous blood will be collected for baseline antibody analysis. Patients will return four weeks later for a follow-up phlebotomy of another 7cc of blood for analysis of functional antipneumococcal antibody generated in response to vaccine antigen challenge. Blood samples will be centrifuged and stored, and stored sera will be sent in batches on dry ice to Flow Applications, Inc. in McDonough, Georgia for antibody analysis. All samples will be assigned unique patient identifiers.

Responses to the 23-valent pneumococcal polysaccharide vaccine will be measured by ELISA to determine the geometric mean increase in immunoglobulin G (IgG) antibody titer to pneumococcal polysaccharide (Pnc Ps) serotypes. Functional antibody, measured by percent kill of a known pneumococcal concentration, will be determined by opsonophagocytosis assay (OPA). Titers for serogroup 4 and serotypes 6B, 19F, and 23F will be measured, and geometric mean rises in antibody concentrations will be determined to measure response to vaccination.

For those treated with nonoperative management, degree of antibody response and grade of splenic injury will be analyzed against normal controls.

Patients treated via splenic artery embolization will undergo a standard post-embolization computed tomographic exam of the abdomen three to five days postinjury to evaluate the effectiveness of the embolization procedure. The percent of viable, perfused spleen will be calculated from this CT. Antibody response will be compared against the location of the intravascular coils (i.e., proximal versus distal embolization) and the percent of viable spleen as calculated on the follow-up CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients (aged 18 to 65 years old) sustaining a splenic injury.

Exclusion Criteria:

* Ages less than 18 and greater than 65
* Initial planned nonoperative management patient who subsequently undergoes embolization or splenectomy will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-12; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Geometric mean increases in pneumococcal antibody titer | 4 weeks
  measured by opsonophagocytosis assay

CONTACTS AND LOCATIONS:
Overall Officials: David Shatz, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/study-of-immune-response-to-pneumococcal-vaccine-in-splenic-injury-patients-999760/